CLINICAL TRIAL: NCT06306638
Title: A Phase I/II Study of Interstitial Photodynamic Therapy Following Palliative Radiotherapy for Patients With Inoperable Malignant Central Airway Obstruction
Brief Title: Interstitial Photodynamic Therapy Following Palliative Radiotherapy in Treating Patients With Inoperable Malignant Central Airway Obstruction
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Modulight, Inc. (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: I-3901323; NCI-2024-01239 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3901323 (Other: Roswell Park Cancer Institute); R01CA283547 (NIH)
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling; Exercise Test; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase I cohort 1 (I-PDT, EBUS) (Experimental): Patients receive visudyne IV over 10 minutes and then undergo I-PDT with EBUS 60-120 minutes after visudyne for up to 3 treatment sessions. Patients undergo blood and tissue sample collection on study. Patients also undergo CT throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Endobronchial Ultrasound Bronchoscopy; Procedure: Interstitial Photodynamic Therapy; Other: Physical Performance Testing; Other: Questionnaire Administration; Drug: Verteporfin
- Phase I cohort 2 (I-PDT, EBUS, palliative radiation therapy) (Experimental): Patients undergo SOC p-XRT over a single fraction. Patients receive visudyne IV over 10 minutes and then undergo I-PDT with EBUS 60-120 minutes after visudyne for up to 2 treatment sessions at least 12 weeks apart. Patients undergo blood and tissue sample collection on study. Patients also undergo CT throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Endobronchial Ultrasound Bronchoscopy; Procedure: Interstitial Photodynamic Therapy; Radiation: Palliative Radiation Therapy; Other: Physical Performance Testing; Other: Questionnaire Administration; Drug: Verteporfin; Device: Laser: ML7710-PDT
- Phase II (I-PDT, EBUS, palliative radiation therapy) (Experimental): Phase II: Patients undergo SOC p-XRT over a single fraction. Patients receive visudyne IV over 10 minutes and then undergo I-PDT with EBUS 60-120 minutes after visudyne for up to 2 treatment sessions at least 12 weeks apart. Patients undergo blood and tissue sample collection on study. Patients also undergo CT throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Endobronchial Ultrasound Bronchoscopy; Procedure: Interstitial Photodynamic Therapy; Radiation: Palliative Radiation Therapy; Other: Physical Performance Testing; Other: Questionnaire Administration; Device: Laser: ML7710-PDT

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Endobronchial Ultrasound Bronchoscopy — Undergo EBUS
  Other Names: EBUS; Endobronchial Ultrasound
Procedure: Interstitial Photodynamic Therapy — Undergo I-PDT
  Other Names: I-PDT; Interstitial Illumination Photodynamic Therapy
Radiation: Palliative Radiation Therapy — Undergo palliative radiation therapy
  Other Names: Palliative Radiotherapy
  Arms: Phase I cohort 2 (I-PDT, EBUS, palliative radiation therapy); Phase II (I-PDT, EBUS, palliative radiation therapy)
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies
Drug: Verteporfin — Given IV
  Other Names: Benzoporphyrin Derivative Monoacid Ring A; BPD-MA; Visudyne
  Arms: Phase I cohort 1 (I-PDT, EBUS); Phase I cohort 2 (I-PDT, EBUS, palliative radiation therapy)
Device: Laser: ML7710-PDT — Delivering the therapeutic 689+/-3 nm laser light during I-PDT. Measuring light transmission.
  Other Names: Fiber-coupled diode laser: ML7710-PDT
  Arms: Phase I cohort 2 (I-PDT, EBUS, palliative radiation therapy); Phase II (I-PDT, EBUS, palliative radiation therapy)

SUMMARY:
This phase I/II trial studies the side effects of interstitial photodynamic therapy following palliative radiotherapy and how well it works in treating patients with inoperable malignant central airway obstruction. Patients who have advanced stage cancer tumors in the lung can often have the breathing passages to the lung partially or completely blocked. These tumors could be due to lung cancer or other cancers (e.g., renal, breast, kidney, etc.) that spread to the lung. This blockage puts the patient at a higher risk for respiratory failure, post-obstructive pneumonia, and prolonged hospitalizations. Treatment for these patients may include bronchoscopic intervention (such as mechanical removal, stenting, laser cauterization, or ballooning), radiation therapy with and without chemotherapy. While palliative x-ray radiotherapy may help in shrinking the tumor, high dose curative radiotherapy that can ablate (a localized, nonsurgical destruction) the tumor also has high risk to cause significant toxicity, including bleeding, abnormal connections or passageways between organs or vessels and abnormal scar tissue that can also produce airway obstruction. Photodynamic therapy (PDT) is another possible treatment that can provide local control of the tumor. PDT consists of injecting a light sensitive drug (photosensitizer, PS) into the vein, waiting for the PS to accumulate in the tumor, and then activating it with a red laser light. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Giving interstitial photodynamic therapy following palliative radiotherapy may improve tumor response and survival without the serious side effects that are associated with the typical high dose curative x-ray radiotherapy alone in patients with malignant central airway obstruction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the safety of our image-based treatment planning for image-guided interstitial photodynamic therapy (I PDT) with endobronchial ultrasound (EBUS) following standard of care palliative radiotherapy (p-XRT). (Phase I)

-To assess the efficacy of our image-based treatment planning for image-guided I-PDT following standard of care p-XRT. (Phase II)

SECONDARY OBJECTIVES:

* To assess objective tumor response. (Phase I)
* To evaluate changes in quality of life. (Phase I and II)
* To measure changes in functional lung capacity. (Phase I and II)
* To measure the relationship between the measured objective tumor response (at 12 +/- 2 weeks post I-PDT) and changes in therapeutic laser light transmission within the target tumor, as a future dosimetric marker for response. (Phase I and II)
* To assess treatment effects on the immune contexture. (Phase I and II)
* To monitor progression free survival. (Phase I and II)

OUTLINE: This is a phase I study, followed by a phase II.

PHASE I: Patients are assigned to 1 of 2 cohorts.

COHORT 1: Patients receive visudyne intravenously (IV) over 10 minutes and then undergo I-PDT with EBUS 60-90 minutes after visudyne for up to 3 treatment sessions. Patients undergo blood and tissue sample collection on study. Patients also undergo computed tomography (CT) throughout the trial.

COHORT 2: Patients undergo SOC p-XRT over a single fraction. Patients receive visudyne IV over 10 minutes and then undergo I-PDT with EBUS 60-90 minutes after visudyne for up to 2 treatment sessions at least 12 weeks apart. Patients undergo blood and tissue sample collection on study. Patients also undergo CT throughout the trial.

PHASE II: Patients undergo SOC p-XRT over a single fraction. Patients receive visudyne IV over 10 minutes and then undergo I-PDT with EBUS 60-90 minutes after visudyne for up to 2 treatment sessions at least 12 weeks apart. Patients undergo blood and tissue sample collection on study. Patients also undergo CT throughout the trial.

After completion of study treatment, patients are followed up at 30 days and 8, 12, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Eligibility checklist before registration requires review of case by the interventional pulmonologist/s and radiation oncologist/s to approve anatomic feasibility of an airway intervention and palliative radiotherapy
* Patients with pathologic diagnosis of inoperable solid malignancy involving extrabronchial tumor growth that causes airway obstruction and not amenable to curative radiotherapy. All patients will have tumors requiring bronchoscopic intervention with endobronchial ultrasound (EBUS) at the time of I-PDT
* Participants have at least one measurable lesion which is also the target lesion for Response Evaluation Criteria in Solid Tumors (RECIST) measurement
* Patients amenable to receive standard of care palliative radiotherapy to the target tumor, as determined by the radiation oncologist/s
* Amenable to high resolution chest CT (with or without contrast due to contraindication) with 0.625-1.25 mm slice thickness and slice interval 0.5-1 mm
* Tumor is accessible and amenable to I-PDT, as determined by the interventional pulmonologist/s
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 3
* Platelets ≥ 100,000 cells/mm^3 (International System of Units [SI] units 100 x 10^9/L)
* International normalized ratio (INR) < 1.5 and activated partial thromboplastin time (aPTT) < 1.5 x ULN. PTT or aPTT per institutional standards for participating external sites
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for 3 months after receiving the study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Pregnant or nursing female participants
* Co-existing ophthalmic disease likely to require slit-lamp examination within the next 30 days following I-PDT treatment
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive the I-PDT
* CT imaging suggestive of target tumor invasion into a major blood vessel (typically proximal to segmental vessels)
* Known hypersensitivity/allergy to porphyrin
* Patients who are not cleared by the anesthesiologist to undergo an advanced bronchoscopy procedure under general anesthesia
* Patients diagnosed with porphyria
* Patients with known allergy to eggs
* Patients unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of >= grade 3 adverse events (Phase I) | Within 30 days post interstitial photodynamic therapy (I-PDT)
  Will will be associated with treatment related adverse events .grade 3 (with attribution of 'possible', 'probable' or 'definite'. Will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v 5.0).
Overall tumor response (Phase II) | At 12 weeks post I-PDT
  Will be assessed by complete response (CR) or partial response (PR) defined by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1) criteria.

SECONDARY OUTCOMES:
Overall tumor response (Phase I) | At 12 weeks post I-PDT
  Will be assessed by CR or PR defined by the RECIST v 1.1 criteria.
Quality of life (Phase I and II) | At study enrollment, immediately prior to p-XRT and I-PDT, and at 4 and 12 weeks
  Will be monitored using the Functional Assessment of Cancer Therapy-Lung. This 36 item self-reported quality of life questionnaire measures responses across six domains: physical well-being, social/family well-being, relationship with doctor, emotional well-being, functional well-being, and additional concerns. This scale was chosen because multiple studies support its validity and use in clinical trials of lung cancer.
Functional lung capacity (Phase I and II) | At study entry (baseline), 30 days and 12 weeks
  Will be measured with the six-minute walk test.
Change in the therapeutic laser light transmission (Phase I and II) | During the I-PDT
  Will be measured with our light dosimetry system.
Association between immune markers and tumor response (Phase I and II) | Prior and 7-10 days after the I-PDT
  will be measured with flow cytometry in fresh blood samples collected prior and 7-10 days after the I-PDT.
Progression free survival (Phase I and II) | Time from date of study treatment to the time of first observed disease progression (RECIST 1.1 criteria) at the treated tumor site or, death due to any cause, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Ivanick, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Abramson Cancer Center, Philadelphia, Pennsylvania